CLINICAL TRIAL: NCT06666478
Title: The Effectiveness of a Specific Exercise Program in Alleviating Work-Related Pain and Improving Mood in Various Occupational Populations
Brief Title: Exercise While at Work Alleviates Work-Related Pain and Improves Mood in Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anastasia Beneka (Other)
Responsible Party: Sponsor-Investigator, Anastasia Beneka, Professor of Physical Rehabilitation, Democritus University of Thrace
Organization: Democritus University of Thrace (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15010/133
Record Dates: First submitted 2024-10-19; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Musculoskeletal Pain
Keywords: exercise at workspace
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise protocol at workspace (Experimental): The exercise protocol at Workspace begins in a sitting position with spinal mobility exercises that mobilize the hips, lumbar spine, thoracic spine, and cervical spine, accompanied by progressive activation of the peripheral joints in the upper limbs. This is followed by multiaxial functional exercises for the trunk and upper limbs, which combine various movements (e.g., lateral bending and twisting) that simulate the positions employees assume while working.
  Subsequently, exercises are performed in an upright position, focusing on stretching and mobilizing the joints and nervous tissue to promote relaxation and release. Coordination, fluid movement, and controlled breathing are emphasized to help workers develop and maintain a stable core while on the job. These principles are essential for workers who are frequently exposed to stressors and physical exertion, as they seek to improve the quality of their movements-namely, smoothness, rhythm, and appropriate speed-while at work.
  Interventions: Other: Exercise protocol at workspace
- Control group (No Intervention): Description: Control group. No exercise intervention. A printed document containing general guidelines for pain management and prevention of pain will be provided, in accordance with international guidelines for non-pharmacological interventions in the prevention of chronic non-specific spinal pain, along with recommended exercises for posture improvement.

INTERVENTIONS:
Other: Exercise protocol at workspace — The exercise protocol at Workspace begins in a sitting position with spinal mobility exercises that mobilize the hips, lumbar spine, thoracic spine, and cervical spine, accompanied by progressive activation of the peripheral joints in the upper limbs. This is followed by multiaxial functional exercises for the trunk and upper limbs, which combine various movements (e.g., lateral bending and twisting) that simulate the positions employees assume while working.
  Subsequently, exercises are performed in an upright position, focusing on stretching and mobilizing the joints and nervous tissue to promote relaxation and release. Coordination, fluid movement, and controlled breathing are emphasized to help workers develop and maintain a stable core while on the job. These principles are essential for workers who are frequently exposed to stressors and physical exertion, as they seek to improve the quality of their movements-namely, smoothness, rhythm, and appropriate speed-while at work.
  Arms: Exercise protocol at workspace

SUMMARY:
The goal of this clinical trial is to learn if specific exercise protocol while at work works to treat musculoskeletal pain such as neck pain, back pain, or shoulders' pain in adults workers. It will also learn about the effectiveness of this exercise protocol in improving their mood while working. The main questions it aims to answer are:

* Does exercise while at work help in alleviating pain due to physical exertion?
* Does exercise while at work help in improving mood in workers? Researchers will compare the exercise group to a control group (no guided exercise during the intervention period) to see if exercise works to treat pain due to physical exertion in various working populations.

Participants will:

* Apply a specific exercise protocol adjusted to their workplace and their job's profile for 2 months with a frequency of 3 times per week
* Fill in questionnaires about their pain, mood state, fatigue scale, functional activities level (SF36), Neck disability Index at the beginning of the study, the end of the study and 2 weeks after the end.

DETAILED DESCRIPTION:
Participants' Inclusion and Exclusion Criteria

The study was announced at a public hospital in Northern Greece and within private companies, as described below. Inclusion criteria required participants to be healthcare employees, office employees (both remote and daily commuting workers), or workers involved in manual cargo handling, heavy industry, or agricultural work. Eligible participants were aged up to 67 years, had more than one year of experience in their current position, and had a diagnosis of work-related nonspecific musculoskeletal pain. Healthcare employees were defined as those working in hospital settings, specifically as surgeons or nurses. Office employees were defined as individuals performing administrative tasks in a seated position, such as secretaries, clerks, or typists.

For the purposes of this study, "nonspecific musculoskeletal pain" was defined as pain that cannot be attributed to fractures, direct trauma, or systemic disease, and for which there is no evidence of root compression requiring surgical treatment.

Description of the Exercise Protocol

The exercise protocol begins in a seated position with spinal mobility exercises that mobilize the hips, lumbar spine, thoracic spine, and cervical spine, alongside progressive activation of the peripheral joints in the upper limbs. This is followed by multiaxial functional exercises for the trunk and upper limbs, incorporating various movements (e.g., lateral bending and twisting) that simulate positions assumed by employees during work tasks.

The subsequent exercises are performed in a standing position, focusing on stretching and mobilizing the joints and nervous tissue to promote relaxation and release. Emphasis is placed on coordination, fluid movement, and controlled breathing to help participants develop and maintain core stability while working. These principles are essential for individuals frequently exposed to physical stressors, enabling them to improve movement quality-specifically, smoothness, rhythm, and appropriate speed-thereby enhancing effectiveness with minimal exertion.

All exercises are conducted with full, rhythmic breathing: inhaling to oxygenate body tissues and exhaling to eliminate cellular waste. At the end of each session, participants engage in a specific diaphragmatic breathing relaxation technique.

Assessment Tools

Visual Analogue Scale (VAS) Pain intensity was assessed using the Visual Analogue Scale (VAS). Using a ruler, the score is determined by measuring the distance in millimeters on a 10-cm line between "no pain" and "severe pain," with a higher score indicating greater pain intensity.

Feeling Scale (FS) The Feeling Scale (FS) is an 11-point bipolar rating scale measuring current mood on a valence dimension. The scale ranges from -5 ("very bad") to +5 ("very good"), with intermediate points such as -3 ("bad"), -1 ("fairly bad"), 0 ("neutral"), +1 ("fairly good"), and +3 ("good").

Fatigue Scale The Fatigue Scale is an 11-item measure that distinguishes between mental fatigue (four items) and physical fatigue (seven items), capturing cognitive difficulties and physical tiredness, respectively. This scale uses a five-point rating system (1 = "never" to 5 = "always") and can produce a total fatigue score. It has demonstrated reliability, validity, and sensitivity to treatment changes.

Greek Modified Neck Disability Index (NDI) The Neck Disability Index (NDI) was used to measure functional disability due to neck pain. Widely regarded as the most valid tool for assessing neck pain-related disability, it consists of 10 questions covering the impact of neck pain on daily activities, including personal care, lifting, reading, working, driving, sleeping, and recreation, as well as on pain itself (e.g., intensity, headache, concentration). Each item is scored from 0 to 5, producing a total score ranging from 0 (no disability) to 50 (maximum disability). Higher scores indicate greater pain and functional disability. The Greek version of the NDI has high validity (Cronbach's alpha: 0.85) and excellent reliability (ICC: 0.93).

36-Item Short Form Health Survey (SF-36) The SF-36 is a widely used questionnaire assessing overall health and quality of life across eight domains: physical functioning, role limitations due to physical health, role limitations due to emotional problems, social functioning, bodily pain, general health perceptions, vitality, and mental health. The SF-36 provides scores for each domain and summary scores for physical and mental health, and is commonly used in both clinical and research settings to evaluate patient-reported outcomes.

Modified Fingertip-to-Floor Distance Test This simple clinical test assesses spinal mobility, particularly in the lower back and hamstrings. The distance between the fingertips and the floor is measured as the participant bends forward as far as possible with knees straight and feet together. This test evaluates flexibility, range of motion, and any movement restrictions.

Lateral Spinal Flexion Lateral Spinal Flexion is a clinical assessment used to measure spinal range of motion during sideways bending. The test evaluates the ability to flex the spine laterally in both directions, helping identify any movement restrictions, imbalances, or asymmetries.

ELIGIBILITY:
Inclusion criteria

* Age 19-67
* experienced either persistent or recurrent pain or discomfort in the neck and/or upper back (back) and/or lower back and/or shoulders at least twice during the three months prior to the start of the study
* The average intensity of pain/discomfort over the last three months, measured on a ten-point numerical pain scale, needed to be between 3-7, where 0 corresponds to "no pain" and 10 corresponds to "unbearable pain."
* Job requiring long hours of sedentary work using computers or other technologies
* Job requiring long hours of bending and lifting weights
* Job requiring long hours in a standing position
* Employment as nurses, doctors, or surgeons
* Manual labor in distribution warehouses
* Manual labor in heavy industry

Exclusion criteria

* significant coexisting respiratory, cardiovascular, vascular, oncological, neoplastic, rheumatological, neurological, or psychiatric disease, severe metabolic disorders, or neuromuscular disorders
* any health issues that prevented them from exercising or had received medical recommendations to exercise only under supervision
* if they were taking prescribed medication or undergoing any treatment (e.g., physical therapy) related to their discomfort in the spine or had another serious orthopedic issue
* individuals with a history of spinal surgery or those who had undergone any other major surgery in the past year
* Those with significant herniated discs, severe scoliosis, severe spondylolisthesis, ankylosing spondylitis, congenital spinal deformities, whiplash injuries, sciatica with pain intensity equal to or greater than that in the lower back, and upper limb pain with intensity equal to or greater than that in the neck were also excluded.
* Individuals with phlebitis or those who were pregnant

Ages: 19 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 980 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | From enrollment to the end of the treatment at 6 weeks and 2 weeks after the end of the treatment
  Visual Analogue Scale (VAS) Pain intensity was assessed using the Visual Analogue Scale (VAS). Using a ruler, the score is determined by measuring the distance in millimeters on a 10-cm line between "no pain" and "severe pain," with a higher score indicating greater pain intensity.
Feeling Scale | From enrollment to the end of the treatment at 6 weeks and 2 weeks after the end of the treatment
  Feeling Scale (FS) The Feeling Scale (FS) is an 11-point bipolar rating scale measuring current mood on a valence dimension. The scale ranges from -5 ("very bad") to +5 ("very good"), with intermediate points such as -3 ("bad"), -1 ("fairly bad"), 0 ("neutral"), +1 ("fairly good"), and +3 ("good").
Neck Disability Index | From enrollment to the end of the treatment at 6 weeks and 2 weeks after the end of the treatment
  The Neck Disability Index (NDI) was used to measure functional disability due to neck pain. Widely regarded as the most valid tool for assessing neck pain-related disability, it consists of 10 questions covering the impact of neck pain on daily activities, including personal care, lifting, reading, working, driving, sleeping, and recreation, as well as on pain itself (e.g., intensity, headache, concentration). Each item is scored from 0 to 5, producing a total score ranging from 0 (no disability) to 50 (maximum disability). Higher scores indicate greater pain and functional disability. The Greek version of the NDI has high validity (Cronbach's alpha: 0.85) and excellent reliability (ICC: 0.93).
Fatigue Scale | From enrollment to the end of the treatment at 6 weeks and 2 weeks after the end of the treatment
  The Fatigue Scale is an 11-item measure that distinguishes between mental fatigue (four items) and physical fatigue (seven items), capturing cognitive difficulties and physical tiredness, respectively. This scale uses a five-point rating system (1 = "never" to 5 = "always") and can produce a total fatigue score. It has demonstrated reliability, validity, and sensitivity to treatment changes.
Short-Form Health Survey 36 - SF-36 | From enrollment to the end of the treatment at 6 weeks and 2 weeks after the end of the treatment
  The SF-36 is a widely used questionnaire assessing overall health and quality of life across eight domains: physical functioning, role limitations due to physical health, role limitations due to emotional problems, social functioning, bodily pain, general health perceptions, vitality, and mental health. The SF-36 provides scores for each domain and summary scores for physical and mental health, and is commonly used in both clinical and research settings to evaluate patient-reported outcomes.
Modified Fingertip-to-Floor Distance Test, Spinal Lateral Flexion | From enrollment to the end of the treatment at 6 weeks and 2 weeks after the end of the treatment
  This simple clinical test assesses spinal mobility, particularly in the lower back and hamstrings. The distance between the fingertips and the floor is measured as the participant bends forward as far as possible with knees straight and feet together. This test evaluates flexibility, range of motion, and any movement restrictions.
Lateral Spinal Flexion Range of Motion | From enrollment to the end of the treatment at 6 weeks and 2 weeks after the end of the treatment
  Lateral Spinal Flexion is a clinical assessment used to measure spinal range of motion during sideways bending. The test evaluates the ability to flex the spine laterally in both directions, helping identify any movement restrictions, imbalances, or asymmetries.

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Gr Beneka, Professor, Principal Investigator — Democritus University of Thrace
Locations (1):
- Department of Physical Education, Sport Science and Occupational Therapy, Komotini, Greece

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared with anybody because of the Companies/Organizations GDPR policy. They are very sensitive with the GDPR.